CLINICAL TRIAL: NCT06553131
Title: Median Versus Ulnar Nerve Quantitative Electromyography Neuromuscular Blockade Monitoring Comparison
Status: Recruiting | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 5240163
Record Dates: First submitted 2024-08-10; First posted 2024-08-14 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Neuromuscular Blockade
Keywords: Median Nerve; Neuromuscular Blockade; Ulnar Nerve

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Surgical Patients Receiving Non-Depolarizing Neuromuscular Blockade: Surgical patients having surgery that requires muscle relaxation with non-depolarizing neuromuscular blockers and monitoring of the depth of muscle blockade.The muscle response to nerve stimulation will be compared between the ulnar and median nerve.
  Interventions: Device: Neuromuscular Transmission Monitoring

INTERVENTIONS:
Device: Neuromuscular Transmission Monitoring — A neuromuscular transmission module connected to electrodes applied to the skin and positioned to provide stimulation of a single nerve and monitor the muscular response to nerve stimulation

SUMMARY:
Medications used to relax the muscles are used during surgery. The amount of muscle relaxation can monitored with devices that stimulate a specific nerve and evaluate the muscle response. The response to, and recovery from, medications that relax the muscles are best described for a nerve in the arm called the ulnar nerve. The investigators believe that other nerves in the arm, such as the median nerve, could be used to monitor the amount of muscle relaxation. The purpose of this study is to compare the muscle response at two different nerve sites after giving medications to relax the muscles.

This study is going to measure the depth of muscle relaxation during surgery at two different sites. The muscle response to stimulation of the ulnar nerve (located in the arm) will be compared to the muscle response to stimulation of the median nerve (also located in the arm).

DETAILED DESCRIPTION:
This is a single-center prospective, randomized controlled trial comparing ulnar versus median nerve electromyography transmission.

Neuromuscular blockade is used to provide muscle relaxation during surgery. The depth of neuromuscular blockade can be monitored with nerve stimulation or electromyography. The response to and recovery from non-depolarizing neuromuscular blockade is best described for the ulnar nerve. The investigators postulate that the median nerve may provide comparable information about the response non-depolarizing neuromuscular blockade. Electromyography electrodes will be positioned to stimulate the ulnar nerve in one arm and the median nerve in the other arm. The response to, and recovery from, non-depolarizing neuromuscular blockade will be compared between the ulnar and median nerve.

The location of median nerve monitoring will be randomized to the dominant or non-dominant hand.

The randomized arm will have electrodes positioned to stimulate the median nerve and the other arm will have electrodes positioned to stimulate the ulnar nerve (standard site for monitoring neuromuscular transmission during anesthesia).

The purpose of the study is to compare the response to, and recovery from, non-depolarizing neuromuscular blockade between the ulnar and median nerves.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 - 75 years of age who are able to provide consent
* Scheduled for elective surgery requiring muscle relaxation, in a supine position under general anesthesia, with an anticipated duration of at least 1.5 hours

Exclusion Criteria:

* Contraindication to rocuronium use
* Comorbidities that may prolong the duration of neuromuscular blockade or alter pharmacodynamics and/or pharmacokinetics, such as:
* Neuromuscular disease
* Expected or known difficult airway
* Rocuronium allergy
* BMI < 18.5 or > 40
* History of adhesive allergy
* Upper extremity weakness, limb deformity, or absence of all or part of an upper limb
* Patients undergoing surgical procedures requiring cardiopulmonary bypass

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery at Loma Linda University Medical Center
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Neuromuscular transmission nerve monitoring concordance | Change in time between administration of rocuronium at beginning of surgery and the appearance of one post-tetanic twitch on a monitor, typically 20 minutes after sedation
  The length of time between rocuronium administration and first post-tetanic twitch for both nerves

SECONDARY OUTCOMES:
Non-inferiority of median nerve neuromuscular monitoring compared to ulnar nerve neuromuscular monitoring - first train of four | Change in time between administration of rocuronium at beginning of surgery and the appearance of the first Train-of-Four twitch on a monitor, typically 30 minutes after appearance of post-tetanic twitch
  Time from rocuronium administration to the patient having 1 Train-of-Four twitch after appearance of first post-tetanic twitch, on both monitors
Non-inferiority of median nerve neuromuscular monitoring compared to ulnar nerve neuromuscular monitoring - second train of four | Change in time between administration of rocuronium at beginning of surgery and the appearance of the first instance of 2 Train-of-Four twitches on a monitor, typically 30 minutes after appearance of first train-of-four twitch
  Time from rocuronium administration to the patient having 2 Train-of-Four twitches after appearance of first Train-of-Four twitch, on both monitors
Non-inferiority of median nerve neuromuscular monitoring compared to ulnar nerve neuromuscular monitoring - reversal | Change in time between administration of sugammadex at end of surgery and the appearance of a Train-of-Four ratio greater than or equal to 0.9 on a monitor, typically 5 minutes after sugammadex administration
  Time from reversal at 2 or more Train-of-Four twitches with sugammadex administration to the patient having a Train-of-Four ratio greater than or equal to 0.9, or 90 percent, on both monitors

CONTACTS AND LOCATIONS:
Overall Officials: Michael Benggon, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Troesch Medical Center, Loma Linda, California, United States

REFERENCES:
- [Background] Iwasaki H, Yamamoto M, Sato H, Doshu-Kajiura A, Kitajima O, Takagi S, Luthe SK, Suzuki T. A Comparison Between the Adductor Pollicis Muscle Using TOF-Watch SX and the Abductor Digiti Minimi Muscle Using TetraGraph in Rocuronium-Induced Neuromuscular Block: A Prospective Observational Study. Anesth Analg. 2022 Aug 1;135(2):370-375. doi: 10.1213/ANE.0000000000005897. Epub 2022 Jan 21. PMID 35061641
- [Background] Ortiz R, Westenberg RF, Langhammer CG, Knaus WJ, Chen NC, Eberlin KR. Nerve Diameter in the Hand: A Cadaveric Study. Plast Reconstr Surg Glob Open. 2019 Mar 13;7(3):e2155. doi: 10.1097/GOX.0000000000002155. eCollection 2019 Mar. PMID 31044121
- [Background] Duvaldestin P, Kuizenga K, Saldien V, Claudius C, Servin F, Klein J, Debaene B, Heeringa M. A randomized, dose-response study of sugammadex given for the reversal of deep rocuronium- or vecuronium-induced neuromuscular blockade under sevoflurane anesthesia. Anesth Analg. 2010 Jan 1;110(1):74-82. doi: 10.1213/ANE.0b013e3181c3be3c. Epub 2009 Nov 21. PMID 19933538
- [Background] Lee HJ, Kim KS, Shim JC, Yoon SW. A comparison of the accuracy of ulnar versus median nerve stimulation for neuromuscular monitoring. Korean J Anesthesiol. 2011 May;60(5):334-8. doi: 10.4097/kjae.2011.60.5.334. Epub 2011 May 31. PMID 21716963
- [Background] Bowdle A, Bussey L, Michaelsen K, Jelacic S, Nair B, Togashi K, Hulvershorn J. A comparison of a prototype electromyograph vs. a mechanomyograph and an acceleromyograph for assessment of neuromuscular blockade. Anaesthesia. 2020 Feb;75(2):187-195. doi: 10.1111/anae.14872. Epub 2019 Oct 16. PMID 31617199